CLINICAL TRIAL: NCT06464536
Title: Tight Surgical Gloves to Prevent Chemotherapy-induced Peripheral Neuropathy: A Randomized Controlled Trial to Evaluate the Efficacy of Compression Therapy in Patients With Taxane-based Chemotherapy for Breast and Urogenital Cancer
Brief Title: Evaluation of the Efficacy of Compression With Tight Surgical Gloves in Patients With Taxane-based Therapy
Acronym: ComPrendo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St.Gallen University of Applied Sciences (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: St.GallenU
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Taxane-induced Peripheral Neuropathy
MeSH Terms: interventions — Gloves, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will wear surgical gloves, patients in the control group will wear gloves of the correct size with a pressure less than 3 mmHg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compression group (Experimental): Participants in the intervention group wear surgical gloves at each taxane administration. The intervention will start 30 minutes before the infusion, continue during the infusion, and last until 30 minutes after the infusion ends. Glove size will be measured on both hands before the first use, following the European standard for medical gloves. The gloves will be worn half a size (0.5) smaller than the appropriate size on both hands. With the help of talcum powder, a second glove of the same size will be worn over the first glove on both hands. After selecting the glove size, the compression strength of the two overlapping gloves will be measured once using a pressure measuring device (PicoPress (c)). The PicoPress(c) device (Microlab Elettronica, Italy) is already in use to measure the pressure of compression bandages. The target range for compression pressure is between 23-32 mmHg (compression class 2) (RAL Deutsches Institut für Gütesicherung und Kennzeichnung e. V., 2008).
  Interventions: Other: Compression
- Control group (Sham Comparator): Participants in the control group will wear two non-compressing surgical gloves of their appropriate size on both hands during each administration of taxanes. The intervention will begin 30 minutes before the infusion, continue during the infusion, and last until 30 minutes after the infusion ends. After selecting the glove size, the compression strength of the two overlapping gloves will be measured once using a pressure measuring device (PicoPress(c)) to verify the pressure. The target range is below 3 mmHg. Measurements with the pressure sensor will be repeated as needed with gloves half a size larger to ensure a low pressure level of less than 3 mmHg.
  Interventions: Other: Compression

INTERVENTIONS:
Other: Compression — conventional surgical gloves that are commonly used in hospitals will be used for compression therapy of both hands
  Other Names: Compression with surgical gloves

SUMMARY:
In this study, the effect of compression therapy of the hands with tight surgical gloves to reduce peripheral neuropathy in adult patients during the application of taxanes will be evaluated.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect of treatment with taxanes. The damage to peripheral nerves leads to pain, numbness, and motor dysfunction, which is very distressing for patients and often results in the reduction of the therapeutic dose of taxanes. Preventive measures are limited, but recent studies show that compression of the hands with tight surgical gloves can significantly reduce the incidence of CIPN. The aim of this randomized controlled trial is to investigate the efficacy of compression therapy in reducing CIPN during taxane-based chemotherapy. The randomized controlled and double-blind study will be conducted at the Comprehensive Cancer Center Zurich (CCCZ) of the University Hospital Zurich from 07/24 to 06/25. Participants will be recruited if they have breast cancer or a urogenital carcinoma and are receiving nab-paclitaxel, paclitaxel, or docetaxel. Exclusion criteria include previous neurotoxic treatment, existing neuropathy, peripheral vascular disease, or the use of medications that affect polyneuropathy. The intervention group will wear surgical gloves with a compression pressure of 23-32 mmHg (equivalent to compression class II) for 30 minutes before, during, and 30 minutes after the infusion. The control group will wear non-compressing gloves with a pressure of less than 3 mmHg. The primary endpoint is the occurrence of moderate to severe CIPN within four therapy cycles, measured according to NCI-CTCAE criteria. Secondary endpoints include patient-reported symptoms and quality of life, assessed by the FACT/COG-NTX questionnaire. Comfort and adherence to the compression therapy will also be evaluated. Participants will be randomized into two groups of 57 each. Data collection and analysis will be conducted according to standardized procedures, and the data will be securely and confidentially stored and managed.

ELIGIBILITY:
Inclusion Criteria:

* Mamma or Urogenital carcinoma
* first treatment with Taxanes (nab-Paclitaxel, Paclitaxel, Docetaxel)
* signed informed consent
* sufficient proficiency in German or English

Exclusion Criteria:

* other therapy that could have caused peripheral neuropathy within the last 24 months (Taxane, Platin, Vincaalkaloids, etc.)
* History of neuropathy such as Raynaud's phenomenon, fibromyalgia and diabetic polyneuropathy
* Use of polyneuropathy medications including duloxetine; gabapentin/pregabalin; topical amitriptyline, ketamine, baclofen; oral cannabinoids; tricyclic antidepressants; and ganglioside monosialic acid
* such impaired cognition that prevents participation in the study according to the assessment of the caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
peripheral polyneuropathy | at the beginning (first day) of each of the first four cycles of chemotherapy for each participant (Cycles range from 7 to 28 days)
  measured with the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grades 0-4 : 0=none, 1=Asymptomatic; clinical or diagnostic observations only, 2=Moderate symptoms; limiting instrumental ADL; 3=Severe symptoms; limiting self care ADL; 4=Life-threatening consequences; urgent intervention indicated (i.e., higher scores meaning worse symptoms)

SECONDARY OUTCOMES:
peripheral polyneuropathy patient reported outcome | at the beginning (first day) of each of the first four cycles of chemotherapy for each participant (Cycles range from 7 to 28 days)
  measured with the neuropathy Subscale of the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group - Neurotoxicity (FACT/COG-NTX), The FACT-NTX subscale comprises 11 5-point ordinal scaled items (0=not at all to 4=very much). The points for each item are totaled and can range from 0=no symptoms to 44=severe symptoms. The participant is counted as a case if the change in the FACT-NTX reaches ≥5 points.
comfort of compression therapy | at the beginning (first day) of each of the first four cycles of chemotherapy for each participant (Cycles range from 7 to 28 days)
  comfort will be measured with a 0 to 3 scale (0=not comfortable at all, 3=very comfortable)
adherence with compression therapy | at the beginning (first day) of each of the first four cycles of chemotherapy for each participant (Cycles range from 7 to 28 days)
  percentage of time that compression should have been administered
Frequency of the application of manual abilities (like sewing, knitting, painting, playing the piano or similar) | at the beginning (first day) of each of the first four cycles of chemotherapy for each participant (Cycles range from 7 to 28 days)
  Ordinal 1-item scale, ranging from from 0=never to 4=daily

CONTACTS AND LOCATIONS:
Overall Officials: Anna Götz, PhD, Principal Investigator — USZ; Antje Koller, PhD, Principal Investigator — St.Gallen University of Applied Sciences
Locations (1):
- University Hospital Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
secondary data analysis are planned to be possible on request, data that may disclose the patients identity will be deleted from the dataset